CLINICAL TRIAL: NCT00316329
Title: Multinational, Randomized, Comparative Study of the Efficacy and Safety of Three Therapeutic Regimens: Coarsucam™ (Artesunate + Amodiaquine Fixed-Dose Combination) Administered in 1 or 2 Intakes Per Day Versus Coartem® (Artemether + Lumefantrine) in the Treatment of Uncomplicated Plasmodium Falciparum Malaria
Brief Title: ATAQ EASY: Artesunate + Amodiaquine Fixed Dose Combination in the Treatment of Uncomplicated Plasmodium Falciparum Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PM_L_0164
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination

INTERVENTIONS:
Drug: Artesunate + Amodiaquine

SUMMARY:
Primary Objective:

* To demonstrate the non-inferiority, in terms of clinical and parasitological efficacy on D28 of administration of Coarsucam™ (artesunate+amodiaquine fixed-dose combination), as a single daily dose, in comparison with administration of Coartem® (artemether+lumefantrine).

Secondary Objectives:

To compare the 3 treatment groups in terms of:

* clinical and parasitological efficacy on D14 and D28 on the global population and on the subpopulation consisting of children aged under 5 years and that for patients aged 5 years and over
* clinical and laboratory safety
* time to parasite clearance
* time to clearance of fever
* changes in gametocytaemia
* impact on anaemia

ELIGIBILITY:
Inclusion criteria:

* adults or children weighing ≥ 10 kg
* residing in the zone covered by the investigating centre throughout the entire follow-up period
* capable of receiving oral treatment
* axillary temperature ≥ 37.5 degrees Celsius at the inclusion visit or history of fever within the previous 24 hours
* infection with Plasmodium falciparum, with parasite density in the blood ranging from 1000 to 200,000 asexual forms per cubic millimetre
* informed consent from each participant or parents (guardians) for the children
* negative urinary pregnancy test for all women of child-bearing age

Exclusion criteria:

* presence of at least one serious or clinical danger sign of malaria: prostration, consciousness disorders, recent and repeated convulsions , respiratory distress, inability to drink, uncontrollable vomiting, macroscopic haemoglobinuria, jaundice, haemorrhagic shock, systolic Blood Pressure < 70 mmHg in adults or < 50 mmHg in children, spontaneous bleeding, inability to sit or stand
* serious concomitant disease
* allergy to one of the investigational medicinal products (drug substance or excipient)
* pregnant women (reported, clinically visible or palpable pregnancy, or positive urinary pregnancy test), or breast-feeding women
* clinically documented heart disease (bradycardia, extrasystoles, exertional dyspnoea, systolic or diastolic extrasystoles, gallop rhythm…)
* history of hepatic and (or) haematological impairment during treatment with amodiaquine
* intake of medication metabolised by cytochrome CYP2D6 (e.g. metoprolol, flecainide, imipramine, amitriptyline, clomipramine) or CYP3A4 (e.g. erythromycin, ketoconazole, itraconazole, cimetidine, HIV protease inhibitors)
* family history of congenital QTc prolongation or sudden death or another clinical condition known to prolong the QTc interval
* intake of medication known to prolong the QTc interval, such as class IA and III antiarrythmics, neuroleptics, antidepressant agents, certain antibiotics including drugs in the macrolide class, fluoroquinolones, imidazole and triazole, antifungal agents, certain non-sedative antihistamines (terfenadine, astemizole) and cisapride
* certain known electrolyte imbalances such as hypokalaemia or hypomagnesaemia
* patient having received artesunate + amodiaquine or artemether + lumefantrine at a suitable dosage within 30 days prior to inclusion

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1032
Dates: Start 2006-03

PRIMARY OUTCOMES:
Clinical and parasitological cure (after PCR correction) on D28 in compliance with WHO classification, for the Coarsucam™ & Coartem® groups

SECONDARY OUTCOMES:
Clinical & parasitological cure (after PCR correction) on D14 & D28 in the global population & in the two subpopulations-Time to clearance of parasitaemia & fever-Changes in gametocytaemia & anaemia during follow-up- Clinical & laboratory safety

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Lameyre, Study Director — Sanofi
Locations (5):
- CHU, Yaoundé, Cameroon
- Centre de santé, Tsiroanomandidy, Madagascar
- Bankoumana, Mali
- Senegal (2):
  - Keur Socé
  - Oussouye

REFERENCES:
- [Derived] Ndiaye JL, Randrianarivelojosia M, Sagara I, Brasseur P, Ndiaye I, Faye B, Randrianasolo L, Ratsimbasoa A, Forlemu D, Moor VA, Traore A, Dicko Y, Dara N, Lameyre V, Diallo M, Djimde A, Same-Ekobo A, Gaye O. Randomized, multicentre assessment of the efficacy and safety of ASAQ--a fixed-dose artesunate-amodiaquine combination therapy in the treatment of uncomplicated Plasmodium falciparum malaria. Malar J. 2009 Jun 8;8:125. doi: 10.1186/1475-2875-8-125. PMID 19505304